CLINICAL TRIAL: NCT01133067
Title: A Prospective Study of Telephonic Contact and Subsequent Physical Follow up of Radically Treated Lung Cancer Patients
Brief Title: Telephonic Contact and Subsequent Physical Follow up Treated Lung Cancer Patients
Acronym: TELE001
Status: Completed | Type: Observational
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, J P AGARWAL, Professor Radiation Oncology, Tata Memorial Hospital
Other Study IDs: PROJECT NO 754
Record Dates: First submitted 2010-05-27; First posted 2010-05-28 (Estimated); Results first posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2017-11

CONDITIONS: Lung Cancer
Keywords: lung cancer; followup; physical follow up; telephonic followup
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Does the routine clinical practice of follow up after primary treatment in lung cancer patients has any utility.

DETAILED DESCRIPTION:
Patients of cancer, after their primary treatment are subsequently called for follow up visits to assess the disease status. This has two important implications from the point of view of resource management. One, patients often have to travel long distances to report to the hospital and have to take care of other logistics such as their accommodation, local travel and food. Further often the patient travels with 1-2 attendants which adds to the logistic burden. Also, these patients of follow up also contribute to the load on existing hospital services. Many authors have speculated that follow-up visits generate anxiety about possible disease recurrence. On the other hand, many others have suggested that although there may be a transient increase in anxiety, patients are ultimately reassured by this practice. Hence, there is no firm evidence for the practice and the need for follow up in oncology care.

ELIGIBILITY:
Inclusion Criteria:

1. All patients of lung cancer treated with a radical aim (e.g surgery, Chemoradiation, surgery followed by adjuvant treatment or any other combination)
2. Patients should have completed radical /adjuvant treatment, if any
3. Patients of both SCLC and NSCLC
4. Patients with at least two telephone numbers (landline/mobile/both)
5. Patients willing to participate

Exclusion Criteria:

1. All patients for palliative intention
2. Patients with less than two contact telephone numbers -

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All curative lung cancer patients after there intial primary treatment who have already been given scheduled appointment shall be called telephonically every 3 months. A set of questions shall be asked to the patient in his /her vernacular during the telephonic interview.After the telephonic interview, the patients shall then report to the cancer care specialist at the Hospital for the due follow up visit.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2010-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: JP AGARWAL, MD, Principal Investigator — Tata Memorial Hospital
Locations (1):
- Tata Memorial Hospital, Mumbai, MS, India

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Total Cohort: Single-arm Prospective cohort
Period: Overall Study
Arm/Group | Total Cohort
Started | 200
Completed | 61
Not Completed | 139
Not completed — Death | 136
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Total Cohort
Number analyzed (Participants) | 200
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 56 [50 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 167
Region of Enrollment [Number; unit: participants]
  India | 200
Stage [Number; unit: participants] — AJCC 7th edition Stage Group
  participants
    Stage I | 20
    Stage II | 25
    Stage III | 152
    Stage IV | 3
Histology [Number; unit: participants]
  Adenocarcinoma | 80
  Squamous Carcinoma | 67
  Other NSCLC | 23
  Small Cell Carcinoma | 30

OUTCOME MEASURES:

1. Primary Outcome: Concurrence Between the Telephonic Interview and the Physician Assessment
Description: The Prevalence and bias adjusted Kappa (PABAK) score for concurrence between telephonic and physician assessment of disease status of each patient at each follow up visit was analysed.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Total Cohort
Number analyzed (Participants) | 200
probability | 0.64 [0.58 to 0.70]

2. Secondary Outcome: Cost Analysis
Description: On average, each patient spent INR 5117.10 on travel and INR 3079.06 on lodging per follow up visit.
Time Frame: 2 years
Population: Patients of lung cancer treated with curative intent and on follow up with our institution
Measure: Mean (Standard Deviation); unit: Indian Rupees
Arm/Group | Total Cohort
Number analyzed (Participants) | 200
Indian Rupees
  Average cost of travel | 5117.10 (10370.91)
  Average cost of lodging | 3079.06 (6929.57)

ADVERSE EVENTS:
Arm/Group | Total Cohort
Serious Adverse Events (participants affected / at risk) | 0/200
Other Adverse Events (participants affected / at risk) | 0/200

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes